CLINICAL TRIAL: NCT03186807
Title: Evaluation of Brain Volume and Dimensions in Healthy Fetuses Using Obstetrics Ultrasound Examination at 14-34 Weeks of Pregnancy.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0564-16
Record Dates: First submitted 2017-06-11; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Normal Fetal Brain Morphology
Keywords: normogram; brain lumination; fetal cortex; ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- low risk pregnancy: Inclusion criteria - Women aged 18-45 years old ,Pregnant women between 14+0 and 34+0 weeks.speaking Hebrew language and eligible for obtaining informed consent.
  Gestation who had a singleton fetus in cephalic presentation, with well documented gestational age by first trimester US scan CRL.
  Biometric measurement within 10th to 90th percentile.and low risk for fetal brain developmental disorders.
  Interventions: Diagnostic Test: ultrasonographic scan of fetal brain

INTERVENTIONS:
Diagnostic Test: ultrasonographic scan of fetal brain — 1. Routine measurement of BPD, HC, OFD, cisterna magna, cerebellum, lateral ventricle(1).
     specific measurements as follow:
  2. Parietoccipital fissures will be measured from the most external border of cortex to the luminar line.
  3. Lateral fissure depths will be measured from the most external border of the insular cortex to the interface confirmed between the subarachnoid space and the skull.
  4. Cingulate fissures will be measured in the mid-coronal plane tracing a perpendicular line from the median longitudinal fissure to the apex of the cingulate fissures.
  6. Calcarine fissures will be measured in the coronal transcerebellar plane as tracing a perpendicular line from the median longitudinal fissure to the apex of the calcarine fissures.

SUMMARY:
The aim of this study is to evaluate the "normal" development of cerebral cortex with quantitative measurement in low risk pregnant women

DETAILED DESCRIPTION:
Study design:

This is a prospective study that evaluates normal fetal brain cortex development from 14 to 34 WG using 2D and 3D ultrasound in singleton low risk pregnancies with unknown obstetrical complications. The clinical and obstetrical data will be obtained prior to the US evaluation; and will include maternal medical and obstetrical data and confirmation of fetal gestational age based on first day of the last menstrual cycle (LMP) supported by well documented CRL from first trimester US. Brain biometric and sulcation analysis includes:

1. Routine measurement of BPD, HC, OFD, cisterna magna, cerebellum, lateral ventricle(1).
2. Parietoccipital fissures will be measured in an axial slice above the transthalamic plane used for the BPD assessment tracing a perpendicular line from the longitudinal fissure to the apex of the parietoccipital fissures (4).
3. Insular depths will be measured in the axial slice located immediately below the anterior commissure and the cavum septum pellucidum, tracing a perpendicular line from the median longitudinal fissure to the most external border of the insular cortex(4).
4. Lateral fissure depths will be measured in the same plane described above, with a continuing line starting from the most external border of the insular cortex to the interface conformed between the subarachnoid space and the skull(4).
5. Cingulate fissures will be measured in the mid-coronal plane tracing a perpendicular line from the median longitudinal fissure to the apex of the cingulate fissures.
6. Calcarine fissures will be measured in the coronal transcerebellar plane as described in ISOUG, tracing a perpendicular line from the median longitudinal fissure to the apex of the calcarine fissures.

Two measurements will be taken by two examiners in order to evaluate intraobserver and interobserver reproducibility.

In all the cases a maximum effort will be undertake to obtain adequate volumes of the brain in order to enable offline evaluation of the different structures.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years old ,Pregnant women between 14+0 and 34+0 weeks.speaking Hebrew language and eligible for obtaining informed consent.

Gestation who had a singleton fetus in cephalic presentation, with well documented gestational age by first trimester US scan CRL.

Biometric measurement within 10th to 90th percentile.

Exclusion Criteria:

* rupture of membranes, severe pre-eclampsia, HELLP syndrome (Hemolysis, elevated liver enzymes, and low platelet count), Twins

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women aged 18-45 years old ,Pregnant women between 14+0 and 34+0 weeks.speaking Hebrew language and eligible for obtaining informed consent.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-06-20 (Estimated); Primary Completion 2019-06-20 (Estimated); Study Completion 2020-06-20 (Estimated)

PRIMARY OUTCOMES:
Cerebral cortex thickness and volume stratified by gestational age | the time required for detailed prenatal ultrasound scan (approximately 60 minute)
  ultrasonographic measurements of fetal cerebral cortex thickness and volume at different gestational age (W/G) (14 W/G - 34 W/G). in order to create normogram and reference values.

IPD SHARING:
Plan to Share IPD: No
This is a prospective study that evaluates normal fetal brain cortex development from 14 to 34 WG using 2D and 3D ultrasound in singleton low risk pregnancies with unknown obstetrical complications. Recruitment at time of visit to our hospital emergency room, outpatient clinic, and hospitalized patient. Each participating women can take part in a single Ultrasonographical scan related to our study objective. The clinical and obstetrical data will be obtained prior to the US evaluation; and will include maternal medical and obstetrical data and confirmation of fetal gestational age based on first day of the last menstrual cycle (LMP) supported by CRL

REFERENCES:
- [Background] Sonographic examination of the fetal central nervous system: guidelines for performing the 'basic examination' and the 'fetal neurosonogram'. Ultrasound Obstet Gynecol. 2007 Jan;29(1):109-116. doi: 10.1002/uog.3909. No abstract available. PMID 17200992
- [Background] Filly RA, Cardoza JD, Goldstein RB, Barkovich AJ. Detection of fetal central nervous system anomalies: a practical level of effort for a routine sonogram. Radiology. 1989 Aug;172(2):403-8. doi: 10.1148/radiology.172.2.2664864.
- [Background] Malinger G, Lerman-Sagie T, Watemberg N, Rotmensch S, Lev D, Glezerman M. A normal second-trimester ultrasound does not exclude intracranial structural pathology. Ultrasound Obstet Gynecol. 2002 Jul;20(1):51-6. doi: 10.1046/j.1469-0705.2002.00743.x. PMID 12100418
- [Background] Egana-Ugrinovic G, Sanz-Cortes M, Figueras F, Bargallo N, Gratacos E. Differences in cortical development assessed by fetal MRI in late-onset intrauterine growth restriction. Am J Obstet Gynecol. 2013 Aug;209(2):126.e1-8. doi: 10.1016/j.ajog.2013.04.008. Epub 2013 Apr 9. PMID 23583839